CLINICAL TRIAL: NCT02238041
Title: An ICU Study of Safety and Accuracy Using the GlucoClear CGM System
Brief Title: GlucoClear ICU Study
Status: Withdrawn | Type: Observational
Why Stopped: Discontinued program
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-02
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Intensive Care Unit Blood Glucose Monitoring
Keywords: Glucose monitoring; Intensive care unit

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GlucoClear System
  Interventions: Device: GlucoClear System

INTERVENTIONS:
Device: GlucoClear System

SUMMARY:
The primary purpose of this Study is evaluation of the safety and accuracy of the GlucoClear CGM System.

DETAILED DESCRIPTION:
Design: Non-randomized, non-treatment, prospective, open label Study.

The GlucoClear System will not display real-time glucose values, glucose trend graphs, or glucose alarms to either the Study subjects or the Study site clinical personnel. There will be no treatment of any subject based on the output of the System.

After providing written informed consent, subjects meeting inclusion/exclusion criteria will be monitored by the System for a maximum of 72 hours.

Up to 51 1 mL blood samples will be drawn from each subject for comparative glucose measurements on blood glucose analyzers over the 72 hour period.

After the GlucoClear Sensor removal, subjects will be contacted for a follow-up assessment 14 days later, and any subsequent adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* 18 years Surgical ICU or surgical ICU plus intermediate care unit stay ≥ 24 hours Signed consent

Exclusion Criteria:

Transplant patient End stage medical conditions or diseases Restricted venous access History of HIT or heparin allergy Contraindication for anti-coagulation Positive pregnancy test In another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an anticipated surgical lCU or surgical lCU plus intermediate care unit stay of at least 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
15/20% Accuracy | During 72 hours of anticipated Sensor dwell time.
  15/20% Accuracy: The proportion of GlucoClear glucose measurements within ± 15 mg/dL of Comparator values < 75 mg/dL and within ± 20% of Comparator values ≥ 75 mg/dL)

SECONDARY OUTCOMES:
12/15% Trend Accuracy | During 72 hours of anticipated Sensor dwell time.
  12/15% Trend Accuracy: The proportion of GlucoClear glu-cose measurements within ± 12 mg/dL of the interpolated value between two sequential Com-parator values if that interpolat-ed comparator value is < 80 mg/dL and within ± 15% of in-terpolated Comparator values ≥ 80 mg/dL).